CLINICAL TRIAL: NCT06484114
Title: A Prospective, Randomized, Double-Blind, Sham-Controlled, Multicenter, Pivotal Study to Assess the Efficacy of Revita® Duodenal Mucosal Resurfacing (DMR) on Body Weight Maintenance in Participants With Obesity and Who Have Achieved at Least 15% Weight Loss on Tirzepatide Obesity Pharmacotherapy
Brief Title: Evaluation of the Safety and Efficacy of Revita® DMR on Body Weight Maintenance in Subjects With Obesity Who Have Achieved at Least 15% Weight Loss on Tirzepatide
Acronym: REMAIN-1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C-00700
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Weight Change Trajectory; Weight Change, Body
Keywords: Weight Management; Obesity; Overweight; Weight; Duodenum; Revita; GLP-1; Tirzepatide; Endoscopic; Weight Maintenance
MeSH Terms: conditions — Obesity; Body-Weight Trajectory; Body Weight Changes; Overweight; Body Weight

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Sham-Controlled, Multicenter
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both the obesity research center team (obesity specialist/endocrinologist, blinded study coordinator, obesity research study staff) and the study participant are blinded to the treatment through the 48-week follow-up visit. The Sponsor (except for unblinded Sponsor personnel [see below]) is blinded to the treatment through the 24-week follow-up visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Training (Other): Sites will gain experience with the study protocol and the Revita DMR procedure in an open-label, single-arm treatment assignment for participants who previously achieved 15% weight loss using a GLP-1
  Interventions: Device: Revita Duodenal Mucosal Resurfacing (DMR)
- Active (Active Comparator): Patients who have achieved >15% weight loss from baseline will receive the Revita DMR Procedure
  Interventions: Device: Revita Duodenal Mucosal Resurfacing (DMR)
- Sham (Sham Comparator): Patients who have achieved >15% weight loss from baseline will receive and endoscopic evaluation and will have a catheter introduced but the Revita DMR procedure will not be performed
  Interventions: Device: Sham

INTERVENTIONS:
Device: Revita Duodenal Mucosal Resurfacing (DMR) — DMR is designed to ablate and re-epithelialize the duodenal mucosal surface, thus allowing nutrients to be exposed to a newly regrown and potentially normalized local mucosa. This implies that the duodenal mucosa surface is abnormal in participants associated with metabolic disorders. The Revita DMR procedure is performed endoscopically with supporting fluoroscopy.
  Arms: Active; Training
Device: Sham — An endoscopic review with non active catheter introduction
  Arms: Sham

SUMMARY:
Fractyl is evaluating Revita Duodenal Mucosal Resurfacing (DMR) in the REMAIN-1 pivotal study, which is designed to include two cohorts - an open label cohort referred to as REVEAL-1, and a randomized cohort, which includes both a midpoint analysis and a pivotal analysis. Patients who previously lost at least 15% of their body weight on a GLP-1 can qualify for the open label REVEAL-1 cohort. The data generated from the REVEAL-1 cohort will be used for open label reporting as the study progresses. The REMAIN-1 randomized cohort will enroll patients living with obesity and a body mass index ("BMI") between 30 and 45 kg/m2 who are not currently on a GLP-1 drug. Patients will be prescribed tirzepatide and titrated to achieve at least 15% total body weight loss, at which time tirzepatide will be discontinued and patients will be randomized to Revita versus sham at 2:1.

Midpoint Analysis of Randomized Cohort:

The midpoint analysis of the randomized cohort will be performed at three months of follow-up on approximately 45 patients, allowing us to assess and report on safety and efficacy signals that could be anticipated in the pivotal analysis. These patients are distinct from those included in the pivotal analysis.

Pivotal Analysis of Randomized Cohort:

The pivotal analysis of the randomized cohort will be performed on approximately 315 patients (distinct from those included in the midpoint analysis) and will evaluate safety and efficacy in the first co-primary endpoint, which is weight regain from the time of tirzepatide discontinuation in Revita DMR versus sham patients at six months, with a primary objective of demonstrating a benefit of Revita DMR versus sham for weight maintenance after GLP-1 discontinuation. The second co-primary endpoint evaluates a responder rate among the Revita DMR treated group at one year to demonstrate the durability of the Revita DMR procedure for weight maintenance after discontinuation of a GLP-1-based therapy.

Secondary objectives will include evaluation of the effectiveness of the Revita DMR procedure on the change in blood glucose levels, cardiovascular disease ("CVD") risk factors, body composition and pre-diabetes status. All patients enrolled in the study will receive diet and lifestyle counseling.

DETAILED DESCRIPTION:
Title A Prospective, Randomized, Double-Blind, Sham-Controlled, Multicenter, Pivotal Study to Assess the Efficacy of Revita® Duodenal Mucosal Resurfacing (DMR) on Body Weight Maintenance in Participants with Obesity Who Have Achieved at Least 15% Weight Loss on GLP-1 Based Pharmacotherapy (REMAIN-1)

Short Title Revita® Duodenal Mucosal Resurfacing for Weight Maintenance (REMAIN-1)

Protocol Number C-00700 Study Population Male and non-pregnant non-lactating females aged 21 -70 years, who do not have type 1 or type 2 diabetes mellitus, and with a body mass index (BMI) ≥ 30 kg/m2 Trial Design Study C-00700 is a multi-Stage study which may be conducted in parallel.

Stage 1 is an open-label training Stage enrolling participants already on GLP-1 based therapy (prior to study enrollment) with at least 15% total body weight loss (TBWL) since initiation of the GLP-1 based drug. Those participants who lost at least 15% total body weight on the GLP-1 based drug and wish to discontinue the use, will be eligible to receive Revita DMR procedure.

An open-label training Stage (Stage 1) will require treating endoscopy sites without prior experience with Revita DMR to perform DMR in up to 4 participants per site prior to treating any participant in the randomization Stage (Stage 2) to ensure consistency of study procedures prior to initiating randomization. Sites with prior Revita DMR training and experience may, but are not required to, enroll participants from this stage in parallel to Stage 2.

Stage 2 is a randomized, double-blind, sham-controlled trial that will investigate the impact of Revita® Duodenal Mucosal Resurfacing (DMR), compared with a sham endoscopic procedure, on the maintenance of body weight loss in participants with obesity (BMI ≥ 30 kg/m2). Eligible participants will receive an open-label, tirzepatide run-in, dose-escalation period of approximately 16-26 weeks duration. Those participants who lose at least 15% total body weight during the tirzepatide run-in treatment period will subsequently discontinue tirzepatide and be randomized to either Revita DMR or a sham procedure.

Randomization at the end of the tirzepatide run-in period for eligible participants will be stratified by sex (male, female) and Baseline BMI (<30 or ≥30 kg/m2).

Stage 2 will consist of two independent Stage parts, Stage 2a and Stage 2b, which will enroll sequentially. Both Stages will enroll, randomize, treat, and follow-up participants in the same manner (DMR vs Sham, 2:1, double blind).

* Stage 2a will consist of approximately 45 randomized participants with a range of 30-60. An exploratory safety and efficacy analysis will be performed after the last participant in Stage 2a completes the 12-week visit or discontinues the study.
* Stage 2b will consist of approximately 315 randomized participants. The final efficacy analysis will be performed after the last participant in Stage 2b completes the 52-week visit or discontinues the study.

Phase Pivotal

Sites/Facilities Multicenter trial with up to 35 Revita treatment centers with experience in advanced endoscopy procedures in the United States

Study Intervention and Sham The Revita® System is an endoscopic treatment consisting of a single catheter and console designed to lift the duodenal mucosa with saline followed by controlled circumferential hydrothermal ablation of the mucosa.

The sham procedure consists of placing the Revita® Catheter into the duodenum for a minimum of 30 minutes with no manipulation of the device or activation of the catheter.

Number of Participants Approximately 865 participants will be screened for the entire study.

Stage 1 (Open-label). Approximately 175 participants will be screened, and up to 100 participants will be treated with Revita DMR.

Stage 2 (Randomized). For Stage 2a, approximately 90 participants will be screened, and approximately 60 participants will be enrolled into the tirzepatide run-in treatment period to successfully randomize approximately 45 participants with a range of 30-60 to DMR or sham in a 2:1 ratio. For Stage 2b, approximately 600 participants will be screened, and approximately 400 participants will be enrolled into the tirzepatide run-in treatment period to successfully randomize approximately 315 participants in a 2:1 DMR (n=210) or sham (n=105) treatment ratio. An upper limit of 75% enrollment of females will be used to ensure a sufficiently large sample of men. No more than 20% of total number of randomized subjects will be treated at any single site.

Study Duration The total estimated time from open enrollment until completion of data analyses is 128 weeks.

Participant Study Duration Stage 1 (Open-Label)

The total participant study duration is approximately 54 weeks in Stage 1 of the study with the following study periods:

* A screening period up to 1 week
* A run-in period:

  * Participants enter the study having already achieved at least a 15% body weight loss on a GLP-1 based drug. After meeting all eligibility criteria in visit 1, participants will go directly to study visit 7, the baseline visit.

Visit 7 (baseline visit): Eligible participants will advance from study visit 1 (screening) immediately to study visit 7 at which time their GLP-1 based drug will be discontinued.

Visit 8 (study intervention): Participants will have study intervention (visit 8) one week after GLP-based drug discontinuation.

For these participants, total participant study duration is approximately 54 weeks.

• Study intervention and follow up: The study intervention and post-study intervention period (52 weeks)-An endoscopic evaluation will first be performed to confirm participant eligibility. Immediately following confirmation of participant eligibility, qualifying participants will receive the DMR intervention. The endoscopy evaluation and study intervention will take place during the same endoscopy session. Post- intervention follow up will occur until 52 weeks after intervention.

Stage 2 (Randomized)

The total participant study duration is approximately 68-78 weeks with the following study periods:

* A screening period up to 1 week
* A tirzepatide run-in dose-escalation period (approximately 16-26 weeks) during which time (and until) participants successfully achieve at least 15% body weight loss.

  * Visit 2-6 (tirzepatide run-in): Tirzepatide will be initiated at the end of visit 2, and dose escalation will occur, as tolerated, during study visits 2-6 up to a maximum tolerated dose as per the tirzepatide FDA approved prescribing information or investigator discretion.
  * Visit 7 (baseline visit): Once at least 15% weight loss is achieved at any of these visits 2-6, participants will immediately advance to study visit 7 as his/her next scheduled study visit. During the interval between the documented ≥ 15% weight loss and study visit 7, participants will continue to abide by the recommended tirzepatide dose-escalation regimen per protocol. At study visit 7, tirzepatide will be discontinued.
  * Visit 8 (study intervention): Participants will have visit 8 one week after tirzepatide discontinuation.

The study intervention and post-study intervention period (52 weeks): An endoscopic evaluation will first be performed to confirm participant eligibility. Immediately following confirmation of participant eligibility, participants will be randomized to receive either the DMR or sham intervention. The endoscopy evaluation and study intervention will take place during the same endoscopy session. Post-study intervention follow up will occur in a blinded manner until 52 weeks after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Participant-provided, written informed consent to participate in the study in accordance with local regulations
2. Adult participants aged 21-70 years, inclusive
3. Prior to tirzepatide therapy, have a BMI of ≥ 30 kg/m2 (obesity) and ≤ 45 kg/m2.
4. Have achieved at least 15% weight loss on tirzepatide therapy at Visit 7 (Participants in Stage 1, who enter the study on tirzepatide, must have a documented pre-tirzepatide weight confirming they have lost at least 15% body weight on tirzepatide)
5. Have a history of at least 1 self-reported, unsuccessful, dietary effort to lose body weight
6. All female participants of childbearing potential must have a negative urine pregnancy test at screening and a negative urine pregnancy test at study visit 7 prior to study intervention. Postmenopausal females with amenorrhea for at least 2 years will be eligible if they are > 50 years of age. Postmenopausal females with amenorrhea for at least 2 years, who are ≤ 50 years, must also have documented serum follicle stimulating hormone levels > 35 mUI/mL
7. Able to walk at least 400 yards (roughly the distance of a track) and climb a flight of stairs without difficulty due to either musculoskeletal injuries/diseases or cardiopulmonary diseases
8. If sexually active, WOCBP must use one of the following birth control methods during the entire course of the study as specified:

   * Intrauterine device in place for at least 3 months before the first dose of tirzepatide and throughout the study
   * Barrier method (condom, diaphragm) with spermicide for at least 14 days before the first dose of tirzepatide and throughout the study
   * Surgical sterilization of the male partner(s) (vasectomy for at least 6 months before first dose of tirzepatide) or
   * Hormonal contraceptives with a barrier method for at least 3 months before the first dose of tirzepatide and throughout the study

Exclusion Criteria:

1. Medical conditions that contraindicate the use of tirzepatide for weight management, as detailed in the tirzepatide prescribing information
2. BMI ≥ 40 kg/m2 at Visit 7
3. Females who are or intend to be pregnant or breastfeeding during the study
4. Known serious hypersensitivity to tirzepatide or any of the excipients in tirzepatide
5. History of infectious liver disease excluding recovered Hepatitis A infection
6. History of pancreatitis within 6 months of screening or any prior history of recurrent pancreatitis (i.e., two or more episodes of pancreatitis)
7. Potentially unreliable participants or those judged by the investigator to be unsuitable for the study
8. Unable or unwilling to follow the dietary restrictions specified by the clinical protocol
9. Known history of or active binge eating disorder or suspected binge eating disorder based on binge eating disorder assessment questionnaire
10. Known history of or active substance abuse including alcohol within the past 2 years that, in the opinion of the investigator, may preclude the participant from following the protocol and completing the study
11. Have history of use of marijuana or tetrahydrocannabinol (THC)-containing products within 3 months of screening or unwillingness to abstain from marijuana or THC-containing products use during the study

    Diabetes-related conditions:
12. History of type 1 or type 2 diabetes (T2D) or screening values consistent with T2D, or history of any genetic form of diabetes
13. HbA1c > 6.5% or fasting glucose > 125 mg/dL consistent with T2D diagnosis according to the American Diabetes Association Standards of Care 2024 (Participants with isolated impaired fasting glucose [100 to 125 mg/dL, inclusive] may enroll in the study)

    Laboratory values or clinical abnormalities:
14. Estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73m2 at screening, as assessed by serum creatinine using the revised 2021 CKD-EPI equation
15. Serum calcitonin level ≥ 20 ng/L at screening if eGFR ≥ 60 mL/min/1.73m2 or serum calcitonin level ≥ 35 ng/L if eGFR < 60 mL/min/1.73m2
16. Fasting triglycerides > 500 mg/dL (> 5.6 mmol/L)
17. Abnormal liver function at screening, defined as any of the following: aspartate aminotransferase (AST) > 3X upper limit of the normal reference range (ULN), ALT > 3X ULN, or serum total bilirubin (TB) > 3X ULN
18. Values of systolic blood pressure (SBP) > 180 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg
19. Any ECG or clinical laboratory abnormality which precludes safe involvement in the study in the opinion of the investigator Gastrointestinal
20. Known structural or functional disorder of the esophagus including any swallowing disorder, esophageal chest pain disorders, drug-refractory esophageal reflux symptoms, or active and uncontrolled GERD defined as Los Angeles Grade C or D esophagitis
21. Known structural or functional disorder of the stomach including active gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (a large hiatal hernia or type II and higher paraoesophageal hernia), cancer, or any other disorder of the stomach
22. Clinically significant gastric-emptying abnormality (i.e., severe gastroparesis or gastric outlet obstruction) including a drug-induced abnormality or an abnormality experienced in a person who chronically takes drugs that directly affect GI motility such as metoclopromide or erythromycin
23. Previous GI surgery to treat the duodenum such as participants who have had a Billroth 2, Roux-en-Y gastric bypass, gastric sleeve, or other similar procedures or conditions
24. Known intestinal autoimmune disease including celiac disease, ulcerative colitis, Crohn's disease, lupus erythematosus, scleroderma, or other autoimmune or connective tissue disorder that affects the small intestine
25. Any history of or current other gastrointestinal condition which would preclude an upper GI endoscopy in the opinion of the investigator Cardiovascular
26. New York Heart Association Class III or IV heart failure within 3 months prior to screening
27. History of myocardial infarction or stroke within 6 months of screening
28. Unstable symptomatic or life-threatening arrhythmia or heart block. Note: Asymptomatic atrial fibrillation is not considered to be life-threatening, and patients with asymptomatic atrial fibrillation will be permitted to enter the study

    Related to other concomitant conditions or medical history:
29. Any concurrent medical condition/disorder or clinically symptomatic cardiovascular, gastrointestinal (including pancreatitis), hematological, pulmonary, psychiatric, acute or chronic infectious disease, active retinal disease or other disorder which, in the investigator's opinion, would interfere with the participant's ability to complete the trial, require administration of treatment that could affect the interpretation of the efficacy or safety variables, or preclude safe involvement in the study
30. Self-reported weight gain > 5 kg within 3 months prior to screening
31. Family history or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia (MEN) syndrome 2
32. History of an active or untreated malignancy or in remission from a clinically significant malignancy within the last 5 years (except for treated basal cell or squamous small cell carcinoma of the skin with no evidence of recurrence)
33. Secondary hypothyroidism or inadequately controlled primary hypothyroidism (thyroid-stimulating hormone [TSH] value outside the range of 0.4 to 6.0 mIU/L at screening)
34. Known thyroid cancer
35. Any uncontrolled endocrine condition such as multiple endocrine neoplasia
36. History of hemoglobinopathies (sickle cell anemia, thalassemia major, sideroblastic anemia) or other blood disorder
37. Any uncontrolled psychiatric disorder as assessed by the investigator
38. Any history of known genetic cause of obesity such as Prader-Willi Syndrome
39. History of COVID infection with prolonged symptoms for >4 weeks

    Related to past or current medication use:
40. Administration of any investigational drug or participation in an interventional clinical research study within 30 days or 5 half-lives (whichever is longer) of screening visit
41. Use of any oral or injectable hypoglycemic agents or any other prescription or over-the-counter diabetes or weight loss medications within 12 months prior to screening visit, (except in the case of tirzepatide use in the stage 1 training arm of the study only)
42. Use of any other medications known to cause weight gain or weight loss in the opinion of the investigator
43. Receiving or have received, within 3 months prior to screening, chronic (>14 days) systemic (excluding inhaled, intraocular, intra-articular or topical) corticosteroid treatment or likely to require (in the opinion of the investigator) concurrent treatment with corticosteroids (excluding inhaled, intraocular, intra-articular or topical) during the course of the study
44. Treatment with antihypertensive or lipid-modifying medications which are not on a stable dose for at least 8 weeks prior to screening or anticipated changes or dose adjustments within 30 days following randomization into the study
45. Treatment with thyroid hormones which are not on a stable dose for at least 8 weeks prior to screening
46. Use of anticoagulation therapy (e.g., warfarin, coumadin, or novel oral anticoagulants [NOACs]) or anti-platelet agents (e.g., thienopyridine) which cannot be discontinued for 5-7 days or 2 drug half-lives before the procedure Other Exclusions
47. Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
48. Fractyl Health employees

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that Revita DMR is superior to sham in percent change in body weight from baseline to week 24 | 24 Weeks
  Percent change in total body weight from baseline to week 24, DMR vs sham
To demonstrate that a majority of Revita DMR participants maintain clinically significant weight loss after discontinuing tirzepatide therapy | 24 weeks
  Percentage of DMR participants who maintain at least 5% total body weight loss from pre-tirzepatide (week -21) to week 24

SECONDARY OUTCOMES:
To demonstrate that Revita DMR is superior to sham in the percent change in body weight, pre-tirzepatide to week 24 post-study intervention | 24 weeks
  Percent change in total body weight from pre-tirzepatide (week -21) to week 24, DMR vs sham
To demonstrate that Revita DMR is superior to sham in the prevention of weight regain following tirzepatide discontinuation and 24 weeks post-study intervention | 24 weeks
  Percentage of participants who maintain at least 10% total body weight loss from pre-tirzepatide (week -21) to week 24, DMR vs sham

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Sullivan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (32):
- United States (32):
  - Helios Clinical Research, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - Hoag Hospital, Newport Beach, California
  - UCLA Santa Monica Medical Center, Santa Monica, California
  - Zenith Clinical Research, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - International Research Associates, Miami, Florida
  - Advent Health, Orlando, Florida
  - K2 Medical Research South Orlando, Orlando, Florida
  - Orlando Health Weight Loss and Bariatric Surgery Institute, Orlando, Florida
  - Synexus Clinical Research Institute - The Villages (AES), The Villages, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Cleveland Clinic, Weston, Weston, Florida
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - American Health Network - Franklin, Franklin, Indiana
  - American Health Network - Greenfield, Greenfield, Indiana
  - Indiana University, Indianapolis, Indiana
  - American Health Network - Muncie, Muncie, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYC Research, Inc. (Endocrine Associates of West Village), Long Island City, New York
  - NYU-Langone, New York, New York
  - Preferred Primary Care Physician Pittsburgh, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physician, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physician, Uniontown, Pennsylvania
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Simcare Medical Research LLC, Sugar Land, Texas
  - University of Washington, Seattle, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No